CLINICAL TRIAL: NCT00229814
Title: Magnetic Resonance Spectroscopic Analysis of Pediatric Tectal Tumors: Insight Into Pathology and Behavior
Brief Title: Study of Brain Tumors (Tectal Tumors) Using Magnetic Resonance Imaging
Status: Withdrawn | Type: Observational
Why Stopped: There were technical difficulties and the study was terminated in 2008
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: Tectal Tumors MRS
Record Dates: First submitted 2005-09-12; First posted 2005-09-30 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Tectal Plate Glioma
Keywords: Tectal Plate Glioma; Tumor; Brain; MRI; Spectroscopy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Tectal plate gliomas are relatively rare tumors of childhood with a reported incidence of 10%. Their typical clinical presentation is symptoms and signs of hydrocephalus and are often incidentally diagnosed in the imaging work-up of children with hydrocephalus. Tectal tumors in children comprise a subcategory of brainstem tumors with unique clinical, imaging, and spectroscopic features. There is debate whether they truly represent brainstem tumors or whether they are a site of benign cellular overgrowth. The majority of these tumors are pathologically benign and show no or minimal growth. Not all tectal plate tumors, however, have this typically benign course. Some can manifest a more aggressive behavior. There have been reports in the past attempting to analyze the histology and behavior of these tumors. None of the prior series looking at these tumors have included Magnetic Resonance Spectroscopy (MRS) analysis.

It is interesting that according to where tumors occur in the brainstem usually indicates what their histology and behavior is. Although not absolute, we know that tumors can have a very poor prognosis versus an extremely good prognosis depending on their location in the brainstem. Yet there are always the cases that do not act in the typical fashion and this is where MRS can prove helpful.

This study is being done to look at a region of the brain, called the tectal plate, in children. This part of the brain can be involved by tumors. Because of the location of the tectal plate, it is usually very difficult and risky to get a biopsy (tissue sample) from this area. Magnetic Resonance Spectroscopy (MRS) is a non-invasive imaging technique that can look at the chemical make up of the brain. MRS may allow us to better understand the nature and behavior of these tumors. However, in order to understand disease in this area, we need to look at the normal chemical make up of the brain in children without tectal plate tumors. Healthy patients are being asked to participate as a normal volunteer. We anticipate having a total of 10 to 12 normal volunteers in the MRS study.

ELIGIBILITY:
Inclusion Criteria:

* patients who are already scheduled for a brain MRI at Children's Healthcare of Atlanta at Scottish Rite for reasons other than tectal plate glioma evaluation

Exclusion Criteria:

* patients with tectal plate glioma

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy volunteer children.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Palasis, M.D., Principal Investigator — Children's Diagnostic Imaging of Atlanta
Locations (1):
- Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia, United States